CLINICAL TRIAL: NCT04172675
Title: A Randomized Phase 2 Study of Erdafitinib Versus Investigator Choice of Intravesical Chemotherapy in Subjects Who Received Bacillus Calmette-Guérin (BCG) and Recurred With High Risk Non-Muscle-Invasive Bladder Cancer (NMIBC) and FGFR Mutations or Fusions
Brief Title: A Study of Erdafitinib Versus Investigator Choice of Intravesical Chemotherapy in Participants Who Received Bacillus Calmette-Guérin (BCG) and Recurred With High Risk Non-Muscle-Invasive Bladder Cancer (NMIBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108699; 42756493BLC2003 (Other: Janssen Research & Development, LLC); 2019-002449-39 (EudraCT Number); 2023-510306-40-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Non muscle invasive bladder cancer (NMIBC); Bacillus calmette- guerin (BCG) failure; BCG unresponsive
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — erdafitinib; Gemcitabine; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Erdafitinib (Experimental): Participants with high-risk non-muscle-invasive bladder cancer (NMIBC) presenting as papillary tumor only (carcinoma in situ [CIS], absent), with disease recurrence after bacillus Calmette- Guerin (BCG) therapy will receive treatment with erdafitinib.
  Interventions: Drug: Erdafitinib
- Cohort 1: Investigators Choice (Active Comparator): Participants with high-risk NMIBC presenting as papillary tumor only (CIS, absent), with disease recurrence after BCG therapy will receive the investigator's choice of either intravesical gemcitabine or intravesical mitomycin C (MMC) or hyperthermic MMC. Participants who are randomized to gemcitabine or MMC or hyperthermic MMC in Cohort 1 and demonstrate a recurrence via investigator disease assessment will have the opportunity to cross over to treatment with erdafitinib.
  Interventions: Drug: Investigator Choice (Gemcitabine); Drug: Investigator Choice (Mitomycin C)
- Cohort 2 (Experimental): Participants with high-risk, BCG- unresponsive NMIBC presenting as CIS with or without concurrent papillary tumor will receive treatment with erdafitinib.
  Interventions: Drug: Erdafitinib
- Cohort 3 (Experimental): Marker lesion study in intermediate-risk NMIBC presenting as papillary disease only. All enrolled participants will receive treatment with erdafitinib.
  Interventions: Drug: Erdafitinib

INTERVENTIONS:
Drug: Erdafitinib — Participants will receive erdafitinib orally beginning on Cycle 1 Day 1 until 2 years of treatment have been completed, disease recurrence, intolerable toxicity, withdrawal of consent, a decision by the investigator to discontinue treatment, or study termination, whichever occurs first. Each cycle is of 28 days.
  Other Names: JNJ-42756493
  Arms: Cohort 1: Erdafitinib; Cohort 2; Cohort 3
Drug: Investigator Choice (Gemcitabine) — Investigator's Choice treatment will be given once weekly for at least 4 doses of induction followed by monthly maintenance for at least 6 months.
  Arms: Cohort 1: Investigators Choice
Drug: Investigator Choice (Mitomycin C) — Investigator's Choice treatment will be given once weekly for at least 4 doses of induction followed by monthly maintenance for at least 6 months.
  Arms: Cohort 1: Investigators Choice

SUMMARY:
The purpose of this study is to evaluate recurrence-free survival (RFS) in participants treated with erdafitinib vs Investigator's Choice, for participants with high-risk non-muscle-invasive bladder cancer (NMIBC) who harbor fibroblast growth factor receptor (FGFR) mutations or fusions, and who recurred after bacillus calmette-guerin (BCG) therapy.

DETAILED DESCRIPTION:
This study enrolls participants with high risk NMIBC and FGFR mutations or fusions. Erdafitinib is an oral pan-fibroblast growth factor receptor (FGFR) 1-4 inhibitor with demonstrated clinical activity in participants with solid tumors, including urothelial carcinoma, with alterations in the FGFR pathway. In Cohort 1, participants will be randomized to erdafitinib or to Investigators Choice (intravesical gemcitabine or intravesical mitomycin C [MMC] or hyperthermic MMC). The study consists of screening period, treatment phase, follow-up phase, and long-term extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, recurrent, non-muscle-invasive urothelial carcinoma of the bladder. Variant pathology are allowed
* Tumor with specified fibroblast growth factor receptor (FGFR) mutations or fusions
* Bacillus Calmette- Guerin (BCG)-unresponsive after adequate BCG therapy or BCG experienced participants
* Refuses or is not eligible for cystectomy (Cohort 1 and Cohort 2 only)
* Eastern Cooperative Oncology Group (ECOG) performance status Grade 0-1
* Must sign an informed consent form (ICF) (or their legally acceptable representative must sign) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* A woman of childbearing potential must have a negative pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) (urine or serum) within 7 days before randomization (Cohort 1) or the first dose of study drug (Cohort 2 and Cohort 3)
* Adequate bone marrow, liver, and renal function as specified in the protocol

Exclusion Criteria:

* Histologically confirmed, muscle-invasive (T2 or higher stage) urothelial carcinoma of the bladder
* Histopathology demonstrating any small cell component, pure adenocarcinoma, pure squamous cell carcinoma, or pure squamous CIS of the bladder
* Prior treatment with an FGFR inhibitor
* Active malignancies other than the disease being treated under study. The only allowed exceptions are: (a) skin cancer treated within the last 24 months that is considered completely cured (b) adequately treated lobular carcinoma in situ (LCIS) and ductal CIS (c) history of localized breast cancer and receiving antihormonal agents, or history of localized prostate cancer (N0M0) and receiving androgen deprivation therapy
* Current central serous retinopathy or retinal pigment epithelial detachment of any grade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (150):
- United States (22):
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - USC Institute of Urology, Los Angeles, California
  - The Urology Center of Colorado, Denver, Colorado
  - Urological Research Network, Hialeah, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Simmons Cancer Institute, Springfield, Illinois
  - University of Kansas, Westwood, Kansas
  - Albany Medical College, Albany, New York
  - NYU Langone Health, New York, New York
  - Great Lakes Physician PC d/b/a Western New York Urology Associates, Sanborn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - The Ohio State University- James Cancer Hospital, Columbus, Ohio
  - Oregon Health And Science University, Portland, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - University of Pittsburgh Medical Center - Cancer Centers, Pittsburgh, Pennsylvania
  - Urology Associates, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin
- Argentina (7):
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, Buenos Aires
  - CEMIC Saavedra, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Centro Urologico Profesor Bengio, Córdoba
  - Hospital Privado de Cordoba, Córdoba
- Australia (4):
  - Flinders Medical Centre, Bedford Park
  - St Vincent s Hospital Sydney, Darlinghurst
  - Macquarie University, Macquarie University
  - Peter MacCallum Cancer Centre, Melbourne
- Belgium (4):
  - AZ Maria Middelares, Ghent
  - UZ Leuven, Leuven
  - CHU Sart-Tilman, Liège
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (14):
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Oncocentro Ceará, Fortaleza
  - Associacao de Combate ao Cancer em Goias - Hospital de Cancer Araujo Jorge, Goiânia
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Nossa Senhora da Conceicao S A, Porto Alegre
  - Instituto de Medicina Integral Professor Fernando Figueira, Recife
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - CEPHO Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Fundacao Faculdade de Medicina Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual IAMSPE, São Paulo
- China (4):
  - Nanjing Drum Tower Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tongji Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
- Czechia (4):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Krajská nemocnice Liberec, Liberec
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
- France (15):
  - Hopital Pellegrin CHU Bordeaux, Bordeaux
  - CHU Gabriel-Montpied, Clermont-Ferrand
  - Hopital Huriez, Lille
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hopital Bichat Claude Bernard, Paris
  - CHU De Poitiers, Poitiers
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Hopital Charles Nicolle, Rouen
  - CHP Saint Gregoire, Saint-Grégoire
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - Centre Hospitalier Universitaire de Nancy - Hôpital Central, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (9):
  - Urologicum Duisburg, Duisburg
  - Klinikum Herne - Urologie, Herne
  - Universitatsklinikum Schleswig Holstein Campus Lubeck, Lübeck
  - Praxisklinik Urologie Rhein/Ruhr - Germany, Mülheim
  - Klinikum rechts der Isar - III. Med. Klinik und Poliklinik, München
  - Universitaetsklinikum Muenster, Münster
  - MVZ Urologie 24 gGmbH, Nuremberg
  - Studienpraxis Urologie Drs. Feyerabend, Nürtingen
  - CUROS - Uberörtliche urologische Gemeinschaftspraxis, Wesseling
- India (6):
  - Health Care Global Enterprises pvt Ltd, Bangalore
  - Rajiv Gandhi Cancer Institute & Research Centre, Delhi
  - King Georges Medical University, Lucknow
  - Meenakshi Mission Hospital and Research Center, Madurai
  - Muljibhai Patel Urological Hospital, Nadiād
  - CIMET s Inamdar Multispeciality Hospital, Pune
- Italy (11):
  - Ente Ecclesiastico Ospedale Generale Regionale F. Miulli, Acquaviva delle Fonti
  - Ospedale Regionale Umberto Parini, Aosta
  - Fondazione Istituto G. Giglio, Cefalù
  - Ospedale Civile di Guastalla, Guastalla
  - Azienda Ospedaliera ''Vito Fazzi'', Lecce
  - UOC Oncologia Ospedale Provinciale di Macerata, Macerata
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Fondazione G Pascale Istituto Nazionale Tumori IRCCS, Napoli
  - Azienda Ospedaliera Sant Andrea, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (16):
  - Juntendo University Hospital, Bunkyō City
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Asahi General Hospital, Chiba
  - Hakodate Goryoukaku Hospital, Hakodate
  - Saitama Medical University International Medical Center, Hidaka
  - Hitachi General Hospital, Hitachi
  - St Marianna University Hospital, Kanagawa
  - Nagoya University Hospital, Nagoya
  - JOHAS Osaka Rosai Hospital, Osaka
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Toranomon Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Fujita Health University Hospital, Toyoake
  - University of Tsukuba Hospital, Tsukuba
  - Yokohama City University Medical Center, Yokohama
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia MCM Krakow, Krakow
  - Uniwersytecki Szpital Kliniczny im. Fryderyka Chopina w Rzeszowie, Rzeszów
  - Samodzielny Publiczny Szpital Kliniczny nr 2 PUM, Szczecin
  - Medical Concierge Centrum Medyczne, Warsaw
  - City Clinic Sp. z o.o., Warsaw
  - Uniwersytecki Szpital Kliniczny, Wroclaw
- South Korea (10):
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Fund. Puigvert, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Instituto Valenciano de Oncologia, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital- Linkou, Taoyuan
- United Kingdom (3):
  - The Christie NHS Foundation Trust Christie Hospital, Manchester
  - Universirty of Sheffield Teaching Hospitals NHS Trust, Sheffield
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Han MA, Maisch P, Jung JH, Hwang JE, Narayan V, Cleves A, Hwang EC, Dahm P. Intravesical gemcitabine for non-muscle invasive bladder cancer. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD009294. doi: 10.1002/14651858.CD009294.pub3. PMID 34125951

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results are presented till final database lock date of 07 August 2024. Cohort 2 and Cohort 3 participants were involved in exploratory efficacy endpoints analysis and thus no efficacy data were reported in outcome measures section for Cohort 2 and 3. With implementation of Protocol Amendment 6 (dated 13 July 2023), long term extension (LTE) phase was added in study.
Groups:
- Cohort 1: Erdafitinib: Participants with high-risk non-muscle-invasive bladder cancer (NMIBC) presenting as papillary tumor only (carcinoma in situ [CIS], absent), with disease recurrence after bacillus Calmette- Guerin (BCG) therapy and who either refused or were not eligible for cystectomy received erdafitinib tablets orally, at a dose of 6 milligrams (mg) once daily starting from Day 1 through Day 28 in each subsequent 28-day cycle starting from Day 1 of Cycle 1 up to disease recurrence or progression, intolerable toxicity, withdrawal of consent, a decision by the investigator to discontinue treatment, or study termination, whichever occurred first (up to 2 years). With the implementation of Protocol Amendment 6 (dated 13 July 2023), participants who benefited from the study drug, as determined by investigator, continued to receive study drug in the LTE phase. The participants who did not enter LTE phase discontinued the study.
- Cohort 1: Investigator's Choice: Participants with high-risk NMIBC presenting as papillary tumor only (CIS, absent), with disease recurrence after BCG therapy and who either refused or were not eligible for cystectomy received the investigator's choice of treatment: either gemcitabine intravesical instillation (4 induction doses: 2000 mg once weekly on Days 1, 8, 15 and 22 of Cycle 1 followed by monthly maintenance dose on Day 1 of Cycle 2 to 7, each cycle of 28 days) or either mitomycin C (MMC) or hyperthermic MMC as an intravesical instillation at the dose of 40 mg/40 milliliter (mL). Additional doses of induction or maintenance were allowed per local standard of care. The choice of drug was determined by the investigator and treatment continued until its completion, disease recurrence, intolerable toxicity, withdrawal of consent, a decision by the investigator to discontinue treatment, or study termination, whichever occurred first (up to 2 years). Participants with locally confirmed high-risk recurrence on Investigator's Choice were offered an option to crossover treatment with erdafitinib until protocol amendment 6 (dated 13 July 2023). With the implementation of Protocol Amendment 6 (dated 13 July 2023), participants who benefited from the study drug, as determined by investigator, continued to receive study drug in the LTE phase. The participants who did not enter LTE phase discontinued the study.
- Cohort 2: Erdafitinib: Participants with high-risk, BCG- unresponsive NMIBC presenting as CIS with or without concurrent papillary tumor and who either refused or were not eligible for cystectomy received erdafitinib tablets orally, at a dose of 6 mg once daily starting from Day 1 through Day 28 in each subsequent 28-day cycle starting from Day 1 of Cycle 1 up to disease recurrence or progression, intolerable toxicity, withdrawal of consent, a decision by the investigator to discontinue treatment, or study termination, whichever occurred first (up to 2 years). With the implementation of Protocol Amendment 6 (dated 13 July 2023), participants who benefited from the study drug, as determined by investigator, continued to receive study drug in the LTE phase. The participants who did not enter LTE phase discontinued the study.
- Cohort 3: Erdafitinib: Participants with intermediate-risk NMIBC presenting as papillary disease only (low grade [Grade 1- Grade 2], Ta or T1, with no previous CIS) received erdafitinib tablets orally, at a dose of 6 mg once daily starting from Day 1 through Day 28 in each subsequent 28-day cycle starting from Day 1 of Cycle 1 up to disease recurrence or progression, intolerable toxicity, withdrawal of consent, a decision by the investigator to discontinue treatment, or study termination, whichever occurred first (up to 2 years). With the implementation of Protocol Amendment 6 (dated 13 July 2023), participants who benefited from the study drug, as determined by investigator, continued to receive study drug in the LTE phase. The participants who did not enter LTE phase discontinued the study.
Period: Overall Study
Arm/Group | Cohort 1: Erdafitinib | Cohort 1: Investigator's Choice | Cohort 2: Erdafitinib | Cohort 3: Erdafitinib
Started | 49 | 24 | 16 | 18
Participants of Cohort 1: Investigator's Choice Crossed Over to Cohort 1 Erdafitinib | 0 | 9 | 0 | 0
Treated | 49 | 23 | 16 | 18
Completed (Participants who died were considered to have completed the study as per protocol.) | 42 | 19 | 15 | 14
Not Completed | 7 | 5 | 1 | 4
Not completed — Withdrawal by Subject | 7 | 5 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Erdafitinib | Cohort 1: Investigator's Choice | Cohort 2: Erdafitinib | Cohort 3: Erdafitinib | Total
Number analyzed (Participants) | 49 | 24 | 16 | 18 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (10.89) | 67 (11.3) | 66.7 (12.37) | 61.6 (9.05) | 66.6 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 2 | 9 | 28
  Male | 37 | 19 | 14 | 9 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 2 | 3 | 19
  Not Hispanic or Latino | 32 | 15 | 11 | 12 | 70
  Unknown or Not Reported | 8 | 4 | 3 | 3 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 14 | 7 | 3 | 1 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 3
  White | 27 | 12 | 9 | 15 | 63
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 3 | 2 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 2 | 3 | 1 | 2 | 8
  Australia | 0 | 0 | 1 | 0 | 1
  Belgium | 1 | 1 | 0 | 0 | 2
  Brazil | 7 | 3 | 1 | 0 | 11
  China | 0 | 2 | 0 | 0 | 2
  France | 5 | 3 | 3 | 1 | 12
  Germany | 2 | 2 | 0 | 0 | 4
  India | 0 | 1 | 0 | 0 | 1
  Italy | 5 | 2 | 1 | 1 | 9
  Japan | 6 | 2 | 3 | 0 | 11
  Poland | 2 | 0 | 1 | 1 | 4
  Korea, South | 8 | 2 | 0 | 0 | 10
  Spain | 2 | 3 | 0 | 0 | 5
  United Kingdom | 3 | 0 | 4 | 3 | 10
  United States | 6 | 0 | 1 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Recurrence-Free Survival (RFS)
Description: RFS was defined as the time from the date of randomization until the date of the reappearance of high-risk disease (high-grade Ta, T1 or carcinoma in situ [CIS]), or death, whichever was reported first. Recurrence was assessed using cystoscopy, bladder mapping, urine cytology, and computed tomography (CT)/ magnetic resonance imaging (MRI) urogram. Participants who were recurrence-free and alive or had unknown status were censored at the last tumor assessment. The Kaplan-Meier method was used to estimate the distribution of overall RFS for each treatment group.
Time Frame: From randomization (Cycle 1 Day 1, pre-dose) up to 48.2 months
Population: Intent-to-Treat (ITT) analysis set included all randomized participants. Participants in Cohort 1 were primarily analyzed by the treatment to which they were assigned, regardless of the actual treatment received. Data for this outcome measure was planned to be collected and analyzed for specified arms only as planned in protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Erdafitinib | Cohort 1: Investigator's Choice
Number analyzed (Participants) | 49 | 24
Months | NA [28.58 to NA] — Here, 'NA' signifies that median and upper limit of 95 percent (%) confidence interval (CI) could not be calculated due to less number of participants with event. | 11.60 [5.29 to NA] — Here, 'NA' signifies that upper limit of 95% CI could not be calculated due to less number of participants with event.
Statistical Analysis 1: Comparison: Cohort 1: Erdafitinib vs Cohort 1: Investigator's Choice; Test type: Superiority; p = 0.0007, Unstratified Log rank; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.13 to 0.61] — Hazard ratio and 95% CI were estimated using a Cox proportional hazards regression model

2. Secondary Outcome: Cohort 1: Recurrence-Free Survival Rate at 6 Months and 12 Months
Description: RFS rate was the proportion of participants who were recurrence-free and alive based on Kaplan-Meier estimates. RFS was defined as the time from the date of randomization until the date of the reappearance of high-risk disease (high-grade Ta, T1 or CIS), or death, whichever was reported first. Recurrence was assessed using cystoscopy, bladder mapping, urine cytology, and CT/ MRI urogram. Participants who were recurrence-free and alive or had unknown status were censored at the last tumor assessment.
Time Frame: At Month 6 and Month 12
Population: ITT analysis set included all randomized participants. Participants in Cohort 1 were primarily analyzed by the treatment to which they were assigned, regardless of the actual treatment received. Data for this outcome measure was planned to be collected and analyzed for specified arms only as planned in protocol.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Cohort 1: Erdafitinib | Cohort 1: Investigator's Choice
Number analyzed (Participants) | 49 | 24
Proportion of participants
  6-month survival rate | 0.96 [0.84 to 0.99] | 0.73 [0.49 to 0.87]
  12-month survival rate | 0.79 [0.64 to 0.89] | 0.44 [0.22 to 0.63]

3. Secondary Outcome: Cohort 1: Time to Progression
Description: Time to progression (TTP) was defined as the time from the date of randomization until the date of first documented evidence of any of the following: disease progression (PD) or death. PD included development of or increase in stage to lamina propria invasion (for example- increase from Ta to T1), development of or increase in stage to muscle-invasive disease (stage greater than or equal to [>=] T2), development of or increase in stage to lymph node (N+) or distant metastasis (M1) disease (participants must have previously been diagnosed with N0 and/or M0 disease), increase in tumor grade from low to high (including CIS).
Time Frame: From randomization (Cycle 1 Day 1, pre-dose) up to 48.2 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Erdafitinib | Cohort 1: Investigator's Choice
Number analyzed (Participants) | 49 | 24
Months | NA [NA to NA] — Here 'NA' signifies that median, lower and upper limit of 95% CI could not be calculated as there were small number of participants with events due to early termination of the participants enrollment. | NA [NA to NA] — Here 'NA' signifies that median, lower and upper limit of 95% CI could not be calculated as there were small number of participants with events due to early termination of the participants enrollment.

4. Secondary Outcome: Cohort 1: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of the participant's death due to any cause.
Time Frame: From randomization (Cycle 1 Day 1, pre-dose) up to 48.2 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Erdafitinib | Cohort 1: Investigator's Choice
Number analyzed (Participants) | 49 | 24
Months | NA [NA to NA] — Here, 'NA' signifies that median, lower and upper limit of 95% CI could not be calculated as there were small number of participants with events due to early termination of the participants enrollment. | NA [NA to NA] — Here, 'NA' signifies that median, lower and upper limit of 95% CI could not be calculated as there were small number of participants with events due to early termination of the participants enrollment.

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs were the events between first dose of study drug and up to 30 (+7 days) days after last dose or before start of subsequent anticancer therapy, whichever occurred first. All TEAEs including serious and non-serious events were reported in this outcome measure (OM).
Time Frame: From start of treatment (Day 1) up to 25.2 months
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Erdafitinib | Cohort 1: Investigator's Choice | Cohort 2: Erdafitinib | Cohort 3: Erdafitinib
Number analyzed (Participants) | 49 | 23 | 16 | 18
Participants | 49 | 19 | 16 | 18

6. Secondary Outcome: Plasma Concentrations of Erdafitinib
Description: Plasma concentrations of erdafitinib were reported. Plasma samples were analyzed using liquid chromatography/mass spectrometry method.
Time Frame: All cohorts: Pre-dose on Cycle 1 Day 14, pre-dose and 3 hours post-dose on Cycle 2 Day 1 (each cycle was of 28 days)
Population: Pharmacokinetic (PK) evaluable analysis set: all randomized (Cohort 1) or treated (Cohort 2 and 3) participants who had received at least 1 dose of erdafitinib and had at least 1 PK sample obtained post-treatment. 'N' (overall number of participants analyzed): number of participants evaluable for this OM, 'n' (number analyzed): participants analyzed at specified time points. Data for this outcome measure was not planned to be collected and analyzed for 'Cohort 1: Investigator's Choice' arm.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Cohort 1: Erdafitinib | Cohort 2: Erdafitinib | Cohort 3: Erdafitinib
Number analyzed (Participants) | 43 | 16 | 18
Nanograms per milliliter (ng/mL)
  Cycle 1 Day 14: Predose: number analyzed (Participants) | 43 | 15 | 18
  Cycle 1 Day 14: Predose | 592 (252) | 525 (227) | 605 (171)
  Cycle 2 Day 1: Predose: number analyzed (Participants) | 43 | 15 | 16
  Cycle 2 Day 1: Predose | 635 (335) | 603 (350) | 685 (246)
  Cycle 2 Day 1: 3 hours post dose: number analyzed (Participants) | 43 | 16 | 12
  Cycle 2 Day 1: 3 hours post dose | 750 (367) | 739 (337) | 709 (220)

ADVERSE EVENTS:
Time Frame: Cohort (C) 1 (Erdafitinib and Investigators Choice), C2 and C3: All cause mortality: From randomization (Cycle 1 Day 1, pre-dose) up to 48.2 months; Serious AEs/Other AEs: From start of treatment (Day 1 of Cycle 1) up to 30(+7 days) days after last dose (up to 25.2 months), C1 crossover participants: All cause mortality: Screening crossover visit (Month 12) up to 48.2 months; Serious AEs/Other AEs: Screening crossover visit (Month 12) up to 30(+7 days) days after last dose (up to 25.2 months)
Description: All cause mortality: analyzed on all randomized participants, Serious AEs (SAEs) and Other AEs: Safety analysis set included all participants who received at least 1 dose of study drug. AEs were collected and analyzed collectively in investigator's arm for gemcitabine or mitomycin C (MMC)/hyperthermic MMC. Per plan safety was analyzed per intervention.
Groups:
- Cohort 1: Crossover Participants From Investigator's Choice to Erdafitinib: Participants in Cohort 1 who initially received investigator's choice of treatment with locally confirmed high-risk recurrence on investigator's choice were offered an option to crossover at crossover screening visit and received erdafitinib tablets orally, at a dose of 6 mg once daily starting from crossover Cycle 1 Day 1 (Month 12) up to disease recurrence or progression, intolerable toxicity, withdrawal of consent, a decision by the investigator to discontinue treatment, or study termination, whichever occurred first (up to 2 years) until protocol amendment 6 (dated 13 July 2023). With the implementation of Protocol Amendment 6 (dated 13 July 2023), participants who benefited from the study drug, as determined by investigator, continued to receive study drug in the LTE phase. The participants who did not enter LTE phase discontinued the study.
Arm/Group | Cohort 1: Erdafitinib | Cohort 1: Investigator's Choice | Cohort 1: Crossover Participants From Investigator's Choice to Erdafitinib | Cohort 2: Erdafitinib | Cohort 3: Erdafitinib
All-Cause Mortality (participants affected / at risk) | 5/49 | 0/24 | 0/9 | 1/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 13/49 | 2/23 | 3/9 | 4/16 | 1/18
Other Adverse Events (participants affected / at risk) | 49/49 | 19/23 | 9/9 | 16/16 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Erdafitinib (N=49) | Cohort 1: Investigator's Choice (N=23) | Cohort 1: Crossover Participants From Investigator's Choice to Erdafitinib (N=9) | Cohort 2: Erdafitinib (N=16) | Cohort 3: Erdafitinib (N=18)
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Central Serous Chorioretinopathy (Eye disorders) | 0 | 0 | 2 | 0 | 0
Detachment of Macular Retinal Pigment Epithelium (Eye disorders) | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Maculopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Enterococcal Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pulmonary Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Brain Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neuroendocrine Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Peripheral Artery Occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Erdafitinib (N=49) | Cohort 1: Investigator's Choice (N=23) | Cohort 1: Crossover Participants From Investigator's Choice to Erdafitinib (N=9) | Cohort 2: Erdafitinib (N=16) | Cohort 3: Erdafitinib (N=18)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Corneal Dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 5 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 2 | 0 | 0 | 3 | 0
Cataract Subcapsular (Eye disorders) | 0 | 0 | 0 | 0 | 1
Central Serous Chorioretinopathy (Eye disorders) | 11 | 0 | 3 | 2 | 2
Corneal Scar (Eye disorders) | 0 | 0 | 0 | 0 | 1
Detachment of Retinal Pigment Epithelium (Eye disorders) | 5 | 0 | 1 | 1 | 2
Dry Age-Related Macular Degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry Eye (Eye disorders) | 11 | 0 | 0 | 4 | 5
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye Pain (Eye disorders) | 2 | 0 | 0 | 0 | 1
Eyelid Oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 2 | 0 | 0 | 1 | 0
Keratopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Lacrimation Increased (Eye disorders) | 8 | 0 | 0 | 2 | 1
Metamorphopsia (Eye disorders) | 0 | 0 | 0 | 0 | 2
Ocular Hyperaemia (Eye disorders) | 3 | 0 | 0 | 1 | 1
Optic Disc Disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 3 | 0 | 0 | 1 | 0
Punctate Keratitis (Eye disorders) | 3 | 1 | 0 | 1 | 2
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal Dystrophy (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal Exudates (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal Vein Occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 0 | 1 | 0 | 0
Serous Retinal Detachment (Eye disorders) | 3 | 0 | 0 | 0 | 0
Subretinal Fluid (Eye disorders) | 1 | 0 | 1 | 1 | 0
Subretinal Hyperreflective Exudation (Eye disorders) | 0 | 0 | 0 | 0 | 1
Swelling of Eyelid (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ulcerative Keratitis (Eye disorders) | 2 | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 3 | 0 | 0 | 1 | 4
Visual Acuity Reduced (Eye disorders) | 2 | 0 | 0 | 1 | 1
Visual Impairment (Eye disorders) | 1 | 0 | 1 | 1 | 1
Vitreous Detachment (Eye disorders) | 1 | 0 | 0 | 0 | 1
Vitreous Floaters (Eye disorders) | 1 | 0 | 0 | 1 | 1
Xerophthalmia (Eye disorders) | 0 | 0 | 1 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 0 | 1 | 1 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Chapped Lips (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 10 | 1 | 1 | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 29 | 3 | 4 | 9 | 15
Dry Mouth (Gastrointestinal disorders) | 23 | 0 | 6 | 9 | 13
Dyspepsia (Gastrointestinal disorders) | 7 | 1 | 2 | 2 | 4
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Faeces Soft (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gingival Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip Blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lip Dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Lip Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 0 | 3 | 5
Oral Dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 22 | 0 | 3 | 8 | 5
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 2
Asthenia (General disorders) | 5 | 0 | 1 | 3 | 4
Enanthema (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 9 | 1 | 2 | 3 | 7
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 1 | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 3 | 2 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0 | 0 | 0
Temperature Intolerance (General disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Balanitis Candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 3 | 0 | 1 | 1 | 2
Covid-19 (Infections and infestations) | 6 | 1 | 0 | 1 | 1
Cystitis (Infections and infestations) | 4 | 2 | 0 | 1 | 0
Eye Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 4 | 1 | 1 | 1 | 1
Nail Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Oral Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 8 | 0 | 0 | 2 | 4
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 9 | 3 | 2 | 5 | 4
Urinary Tract Infection Bacterial (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Injury Corneal (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 6 | 2 | 1 | 5 | 3
Aspartate Aminotransferase Increased (Investigations) | 6 | 3 | 1 | 3 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 1 | 0 | 0 | 1
Blood Calcium Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 2 | 0 | 0 | 1 | 1
Blood Parathyroid Hormone Increased (Investigations) | 1 | 0 | 0 | 1 | 1
Blood Phosphorus Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Phosphorus Increased (Investigations) | 2 | 0 | 0 | 1 | 1
Cardiac Murmur (Investigations) | 0 | 0 | 0 | 0 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 1 | 0 | 1 | 0
Intraocular Pressure Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Lipase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Ophthalmological Examination Abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 7 | 0 | 0 | 5 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 11 | 0 | 2 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 36 | 0 | 6 | 9 | 18
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0 | 0
Bone Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 2 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 2 | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 1 | 1
Dysgeusia (Nervous system disorders) | 11 | 0 | 0 | 7 | 10
Headache (Nervous system disorders) | 2 | 2 | 0 | 1 | 4
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 0 | 0 | 2 | 2
Taste Disorder (Nervous system disorders) | 2 | 0 | 1 | 0 | 2
Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 4 | 2
Libido Decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 3 | 3 | 1 | 3 | 2
Haematuria (Renal and urinary disorders) | 1 | 3 | 0 | 4 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 0 | 2 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Strangury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Epididymal Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Genital Lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Penile Erosion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Scrotal Dermatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Testicular Atrophy (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0 | 2
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 2 | 0 | 4
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 2 | 6
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 0 | 2 | 3 | 6
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 12 | 0 | 3 | 7 | 9
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hair Texture Abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0 | 1
Nail Bed Inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 2 | 2
Nail Disorder (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 6 | 5
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 16 | 0 | 3 | 2 | 4
Nail Hypertrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Nail Toxicity (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 10 | 0 | 0 | 3 | 5
Onychomadesis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 6 | 0 | 0 | 5 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 4 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 4 | 1
Hypotension (Vascular disorders) | 3 | 0 | 0 | 0 | 0
Superficial Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Varicose Vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04172675/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT04172675/SAP_001.pdf